CLINICAL TRIAL: NCT05415930
Title: Evaluation of an Adaptative, Multidisciplinary, Reach-out Program, Facilitating Pre Exposition
Brief Title: Evaluation of an Adaptative, Multidisciplinary, Reach-out Program, Facilitating Pre Exposition HIV Prophylaxis (PrEP) Prescription and Retention in Care, in a Group of Trans Womens (TW) at High Risk of HIV Infection.
Acronym: PrEP à porter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Other Study IDs: IMEA 066
Record Dates: First submitted 2022-04-20; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-04

CONDITIONS: Transgenderism
MeSH Terms: conditions — Transsexualism | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychosocial assistance — Firs evaluation at Acceptess-T locals by a health mediator specialised in transidentity : advice for administrative procedures (health insurance, residency permit, housing, etc.) management of others social issues Orientation to Acceptess-T sexual health space for medical evaluation Orientation to Acceptess-T mental health space if needed : special focus on sexual health and gender related issues
Other: Medical care — Sexual health clinics at Acceptess-T health space First STI risk evaluation: HIV, HCV, HBV, syphilis TROD realisation Spanish speaking Infectious Diseases (ID) specialist (from ID Department of Bichat hospital) first evaluation Proposition of PrEP if indicated Orientation for hospital follow-up in dedicate PrEP clinics Prescription and follow-up of a feminazing hormonal therapy if needed
Other: Legal-Administrative Assistance — Legal counselling, provided by a sex worker union representative Access to FAST (fond action social trans) which give an economic help to TW in high precarity situations
Other: Focus Group — A group of 10-15 TW, identified through convenience sampling, along with the Acceptess-T "Health Space" multidisciplinary team will be invited to participate in an Human Centered Design (HCD) project.
  The project will be led by a team of anthropologists and sociologists and exchanges will be recorded and fully transcribed and analysed by a person competent in qualitative methodology.
  The objective will be to co-create tailored solutions that meet the needs of TW and are viable to implement within the health system, so TW can be better managed The solutions ideated will work synergistically towards improving TW PrEP access and adherence and health system retention.This is an adaptative program : if new solutions to face PrEP barriers are created during the study follow-up, new mesures will be added to the intervention.

SUMMARY:
Evaluation of an adaptative, multidisciplinary, reach-out program, facilitating pre exposition HIV prophylaxis (PrEP) prescription and retention in care, in a group of trans womens (TW) at high risk of HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Trans woman ≥ 18 years old; Negative HIV-1 and HIV-2 serology; Participant on PrEP or request to start PrEP or reporting present, past or future exposure to HIV; Participant agreed with the constraints imposed by the study (every 3 months visits); Non opposition.

Exclusion Criteria:

* Subject with positive HIV serology; Subject with clinical signs suggesting a primary HIV infection; Subjects planning to travel/live abroad for more than 3 consecutive months or planning to live outside Ile-de-France region; Creatinine clearance < 60 mL/min (Cockroft's formula); History of chronic kidney disease, osteoporosis, osteopenia; Subject receiving a potentially nephrotoxic treatment (long-term nonsteroidal anti-inflammatory drugs); Ongoing post-exposure antiretroviral therapy (the participant may be tested 6 weeks after the end of treatment); Treatment under investigation; Chronic gastrointestinal illness (or chronic nausea or vomiting) interfering with intestinal absorption; HBs antigen positive or with an isolated anti-HBc antibody if participant is not ready to take continuous PrEP; Life-threatening illness (cancer) or other serious illness (cardiovascular, renal, pulmonary, unstable diabetes) which would require treatment that could interfere with treatment adherence; Hypersensitivity to one of the components of TDF / FTC.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trans woman , Negative HIV-1 and HIV-2 serology; Participant on PrEP or request to start PrEP or reporting present, past or future exposure to HIV;
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is the healthcare retention rate over the first 48 weeks study. | 48 weeks
Primary endpoint is the healthcare retention rate over the 96 weeks study. | 96 weeks

SECONDARY OUTCOMES:
1. Total number of TW followed-up for PrEP in the Infectious Diseases Department of Bichat Hospital at W48 | Weeks 48
2. Total number of TW followed-up for PrEP in the Infectious Diseases Department of Bichat Hospital at W96. | Weeks 96
Epidemiological and clinical data assessment. | Week 96
3. PrEP adherence questionnaire at W-4 | Week- 4
3. PrEP adherence questionnaire at Week 4 | Week 4
3. PrEP adherence questionnaire at Week 12 | Week 12
3. PrEP adherence questionnaire at Week 24 | Week 24
3. PrEP adherence questionnaire at Week 48 | Week 48
3. PrEP adherence questionnaire at Week 96 | Week 96
Incidence of clinical and laboratory adverse events or those leading to discontinuation of PrEP from W4 to W96. | Week 96
Concomitant treatment (including hormonal therapy) from W-4 to W96. | Week 96
Number of HIV seroconversion from D1 to W96. | Week 96
Incidence of sexually transmitted infections from D1 to W96.participants | week 96
8. Questionnaire to explore PrEP barriers, difficulties and expectations of study participants from W-4 to W96. | Week -4
Questionnaire to explore PrEP barriers, difficulties and expectations of study participants from W-4 to W96. | Week 24
Questionnaire to explore PrEP barriers, difficulties and expectations of study participants from W-4 to W96. | Week 48
Questionnaire to explore PrEP barriers, difficulties and expectations of study participants from W-4 to W96. | Week 96
Precariousness score from W-4 to W96 | Week -4
Precariousness score from W-4 to W96 | Day 1
Precariousness score from W-4 to W96 | Week 24
Precariousness score from W-4 to W96 | Week 48
Precariousness score from W-4 to W96 | Week 96
Multi modal intervention compliance from D1 to W96 | Week 96
Satisfaction questionnaire from D1 to W96 | Day 1
Satisfaction questionnaire from D1 to W96 | Week 12
Satisfaction questionnaire from D1 to W96 | Week 24
Satisfaction questionnaire from D1 to W96 | Week 48
Satisfaction questionnaire from D1 to W96 | Week 96
Global quality of life questionnaire from W-4 to W96. | Week-4
Global quality of life questionnaire from W-4 to W96. | Day1
Global quality of life questionnaire from W-4 to W96. | Week 24
Global quality of life questionnaire from W-4 to W96. | Week 48
Global quality of life questionnaire from W-4 to W96. | Week 96

IPD SHARING:
Plan to Share IPD: No